CLINICAL TRIAL: NCT01606436
Title: A Placebo- and Positive-Controlled Study of the Electrophysiological Effects on the QT Interval After a Supratherapeutic Dose of LY2140023 in Subjects With Schizophrenia
Brief Title: A Study Measuring Effect of LY2140023 (Pomaglumetad Methionil) on Electrocardiographs in Participants With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 12676; H8Y-MC-HBCG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2012-09

CONDITIONS: Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia | interventions — LY 2140023; pomaglumetad methionil; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 400 mg LY2140023 (Experimental): 400 milligrams (mg) LY2140023 (5 x 80 mg tablets) administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
  Interventions: Drug: LY2140023
- Placebo (Placebo Comparator): Placebo tablets (5) matching LY2140023 administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
  Interventions: Drug: Placebo
- 400 mg Moxifloxacin (Other): Positive control, unblinded 400 milligrams (mg) moxifloxacin (1 x 400 mg tablet) administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: LY2140023 — Administered orally.
  Other Names: pomaglumetad methionil
  Arms: 400 mg LY2140023
Drug: Placebo — Administered orally.
  Arms: Placebo
Drug: Moxifloxacin — Administered orally.
  Other Names: Avelox
  Arms: 400 mg Moxifloxacin

SUMMARY:
This study determined if a single dose of LY2140023 (pomaglumetad methionil) affects the electrical activity in the heart in participants with schizophrenia. This study also helped determine how a single high dose of LY2140023 is tolerated by participants.

DETAILED DESCRIPTION:
The primary objective of this study was to determine that a single supratherapeutic dose of LY2140023 does not differ from placebo in the mean change from baseline in 12-lead electrocardiogram (ECG) QT interval measurements, such that the upper bound of the 2-sided 90% confidence interval (CI) for the greatest time-matched mean effect is <10 ms in subjects with schizophrenia. The secondary objective was to further evaluate the tolerability of a supratherapeutic single dose of LY2140023 monohydrate.

Male or female subjects diagnosed with schizophrenia and aged between 18 and 65 years, inclusive, who had not been hospitalized for psychiatric illness for at least 12 weeks prior to Day 1 of the lead-in period, and who had a Clinical Global Impression - Severity scale score of <4 were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Female participants who are postmenopausal
* Not hospitalized for psychiatric illness for at least 12 weeks prior to Day 1 of the study and have a Clinical Global Impression Severity Scale score of <4
* Willing and able to be hospitalized from Day 1 to the end of the study
* Can be washed out of their antipsychotic medication for the duration of the study
* Considered reliable, able to understand, and willing to perform all study procedures
* Understand the nature of the study and give written informed consent
* Clinical laboratory test results within normal reference range
* Venous access sufficient to allow blood sampling
* Clinically acceptable sitting blood pressure and heart rate

Exclusion Criteria:

* Currently enrolled in, have completed or have discontinued from a clinical trial involving an investigational drug within the last 30 days
* Known allergies to pomaglumetad methionil (LY2140023) or its active metabolite (LY404039), moxifloxacin, related compounds, or components
* Previously completed this study or prematurely discontinued from any study after having received at least 1 dose of pomaglumetad methionil (LY2140023)
* Received treatment with clozapine
* Received aripiprazole within 2 months prior to screening
* Taking either thioridazine or thiothixene
* Receiving treatment with depot antipsychotic medication within 12 weeks, prior to screening
* Taking any medications other than those that are specifically permitted in the protocol
* Asthma needing active beta 2 (B2) agonist within 14 days of the study
* Active suicidal ideation with some intent to act, without specific plan or with specific plan and intent or had suicidal behavior such as actual attempt, interrupted attempt, aborted attempt, preparatory act, or behavior within the past 3 months
* Substance dependence or substance abuse (except nicotine and caffeine) within the 6 months prior to admission
* Substance-induced psychosis within 7 days of admission (or at any time during the dosing period)
* History of 1 or more seizures (with exceptions)
* Screening electroencephalogram (EEG) with paroxysmal (epileptiform) activity
* Have had electroconvulsive therapy (ECT) within 3 months of Day 1 of the study or who are expected to have ECT at any time during the live phase of this study
* Parkinson's disease, dementia-related psychosis, or related disorders
* Untreated hyperthyroidism or hypothyroidism needing a thyroid hormone supplement who have not been on a stable dose of medication for at least 2 months prior to screening
* History of leukopenia or agranulocytosis
* Alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) or aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) values greater than 2 times the upper limit of normal (ULN) or total bilirubin values greater than 1.5 times the ULN of the performing laboratory at screening
* Abnormality in the 12-lead electrocardiogram (ECG) that increases the risks associated with participating in the study
* Premature ventricular contraction (PVC) associated with symptoms and/or any complex PVCs
* Heart rhythm disturbance by history or ECG at screening
* Personal or family history of long QT wave syndrome
* Family history of sudden unexplained death or cardiac death in a family member under 60 years of age
* Unexplained syncope within the last year
* Acute, serious, or unstable medical conditions
* Prolactin level of greater than 200 nanograms per milliliter (ng/mL) (200 micrograms per liter [ug/L] or 4228 milli-international units per liter [mIU/L]) at screening (with the exception of participants treated with risperidone) at screening
* Medical history of Human Immunodeficiency Virus positive (HIV+) status
* Test positive for (1) Hepatitis C virus antibody or (2) Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody
* Smoke greater than or equal to 40 cigarettes per day
* Movement disorder that could interfere with conducting 12-lead ECGs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants had to go through a lead in 7-day antipsychotic medication washout.
Groups:
- LY2140023 Then Placebo Then Moxifloxacin: Single 400-mg oral dose of LY2140023 - Day 8 Washout - Days 9-10 Single oral dose of LY2140023-matched placebo - Day 11 Washout - Day 12-13 Single 400-mg oral dose of moxifloxacin (Avelox) - Day 14 Washout - Day 15-16
- Placebo Then Moxifloxacin Then LY2140023: Single oral dose of LY2140023-matched placebo- Day 8 Washout - Days 9-10 Single 400-mg oral dose of moxifloxacin (Avelox)- Day 11 Washout - Day 12-13 Single 400-mg oral dose of LY2140023 - Day 14 Washout - Day 15-16
- Moxifloxacin Then LY2140023 Then Placebo: Single 400-mg oral dose of moxifloxacin (Avelox)- Day 8 Washout - Day 9-10 Single 400-mg oral dose of LY2140023 - Day 11 Washout - Day 12-13 Single oral dose of LY2140023-matched placebo- Day 14 Washout - Days 15-16
- Placebo Then LY2140023 Then Moxifloxacin: Single 400-mg oral dose of placebo- Day 8 Washout - Day 9-10 Single 400-mg oral dose of LY2140023- Day 11 Washout - Day 12-13 Single oral dose of moxifloxacin (Avelox) - Day 14 Washout - Days 15-16
- Moxifloxacin the Placebo Then LY2140023: Single oral dose of moxifloxacin (Avelox) - Day 8 Washout - Day 9-10 Single 400-mg oral dose of placebo- Day 11 Washout - Day 12-13 Single 400-mg oral dose of LY2140023- Day 14 Washout - Days 15-16
- LY2140023the Moxifloxacin the Placebo: Single 400-mg oral dose of LY2140023- Day 8 Washout - Day 9-10 Single oral dose of moxifloxacin (Avelox) - Day 11 Washout - Day 12-13 Single 400-mg oral dose of placebo- Day 14 Washout - Days 15-16
Period: Overall Study
Arm/Group | LY2140023 Then Placebo Then Moxifloxacin | Placebo Then Moxifloxacin Then LY2140023 | Moxifloxacin Then LY2140023 Then Placebo | Placebo Then LY2140023 Then Moxifloxacin | Moxifloxacin the Placebo Then LY2140023 | LY2140023the Moxifloxacin the Placebo
Started | 14 | 14 | 14 | 14 | 13 | 14
Received First Intervention | 14 | 14 | 14 | 14 | 13 | 14
Received Second Intervention | 14 | 14 | 14 | 14 | 12 | 14
Received Third Intervention | 14 | 14 | 12 | 12 | 12 | 14
Completed | 14 | 14 | 12 | 12 | 12 | 14
Not Completed | 0 | 0 | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Overall: After completing a 7-day antipsychotic medication washout period (Days 1 to 7), participants still meeting eligibility criteria were randomized to receive single doses of LY2140023 (Treatment A), matching placebo (Treatment B), and moxifloxacin (Treatment C) in 1 of 6 treatment sequences (ABC, BCA, CAB, BAC, CBA, or ACB). Study drug was administered on Days 8, 11, and 14 of the study.
  LY2140023 (pomaglumetad methionil): 400 milligrams (mg) (5 x 80 mg tablets), administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
  placebo: 5 tablets, administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
  moxifloxacin: 400 mg tablet, administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
Arm/Group | Overall
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 84
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2
  Black or African American | 65
  Native Hawaiian or Other Pacific Islander | 2
  White | 17
Region of Enrollment [Number; unit: participants]
  United States | 86
Weight [Mean (Standard Deviation); unit: kilograms] | 86.73 (15.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline up to 12 Hours Postdose in QT Interval Corrected for Heart Rate (QTc)
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave. QT intervals from quadruplicate electrocardiogram (ECG) data were corrected for heart rate using Fridericia's formula: QTcF = QT/RR^0.333, where RR is the interval between two R waves. Least squares (LS) mean changes from baseline in QTcF were calculated using a mixed-effects model with baseline QTcF, treatment, time, period, sequence, and the time-by-treatment interaction as fixed effects and participant and the participant-by-period interaction as random effects.
Time Frame: Baseline, up to 12 hours postdose in each treatment period
Population: All participants who received at least 1 dose of LY2140023, moxifloxacin, or placebo and had evaluable QTcF data
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- 400 mg LY2140023: LY2140023 (pomaglumetad methionil): 400 milligrams (mg) (5 x 80 mg tablets), administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
- 400 mg Moxifloxacin: moxifloxacin: 400 mg tablet, administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
- Placebo: placebo: 5 tablets, administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
Arm/Group | 400 mg LY2140023 | 400 mg Moxifloxacin | Placebo
Number analyzed (Participants) | 81 | 82 | 80
milliseconds
  0.5 hours: number analyzed (Participants) | 79 | 80 | 79
  0.5 hours | -7.1 [-8.5 to -5.6] | -6.66 [-8.21 to -5.11] | -7.7 [-9.2 to -6.2]
  2.0 hours: number analyzed (Participants) | 76 | 80 | 79
  2.0 hours | -4.7 [-6.2 to -3.2] | -2.62 [-4.18 to -1.07] | -7.6 [-9.1 to -6.1]
  3.0 hours: number analyzed (Participants) | 76 | 81 | 79
  3.0 hours | -4.0 [-5.5 to -2.5] | 0.23 [-1.32 to 1.77] | -6.1 [-7.5 to -4.6]
  4.0 hours: number analyzed (Participants) | 75 | 81 | 79
  4.0 hours | -1.4 [-2.9 to 0.2] | 3.52 [1.98 to 5.07] | -2.8 [-4.3 to -1.4]
  5.0 hours: number analyzed (Participants) | 75 | 0 | 79
  5.0 hours | -2.0 [-3.5 to -0.5] |  | -3.5 [-5.0 to -2.0]
  6.0 hours: number analyzed (Participants) | 76 | 0 | 78
  6.0 hours | -2.6 [-4.1 to -1.1] |  | -6.1 [-7.6 to -4.6]
  8.0 hours: number analyzed (Participants) | 76 | 0 | 76
  8.0 hours | -5.8 [-7.3 to -4.3] |  | -7.9 [-9.4 to -6.4]
  12.0 hours: number analyzed (Participants) | 76 | 79 | 78
  12.0 hours | -6.3 [-7.8 to -4.8] | -3.25 [-4.81 to -1.69] | -8.0 [-9.5 to -6.5]
Statistical Analysis 1: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 0.5 hours postdose; Test type: Superiority or Other; LS Mean Difference = 0.62, 90% CI 2-sided [-1.20 to 2.44]
Statistical Analysis 2: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 2.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 2.89, 90% CI 2-sided [1.05 to 4.73]
Statistical Analysis 3: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 3.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 2.11, 90% CI 2-sided [0.28 to 3.95]
Statistical Analysis 4: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 4.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 1.48, 90% CI 2-sided [-0.36 to 3.32]
Statistical Analysis 5: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 5.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 1.48, 90% CI 2-sided [-0.36 to 3.32]
Statistical Analysis 6: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 6.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 3.48, 90% CI 2-sided [1.64 to 5.32]
Statistical Analysis 7: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 8.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 2.12, 90% CI 2-sided [0.27 to 3.97]
Statistical Analysis 8: Comparison: 400 mg LY2140023 vs Placebo; Comparison at 12.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 1.67, 90% CI 2-sided [-0.17 to 3.51]
Statistical Analysis 9: Comparison: 400 mg Moxifloxacin vs Placebo; Comparison at 0.5 hours postdose; Test type: Superiority or Other; LS Mean Difference = 1.01, 90% CI 2-sided [-1.57 to 3.59]
Statistical Analysis 10: Comparison: 400 mg Moxifloxacin vs Placebo; Comparison at 2.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 4.99, 90% CI 2-sided [2.40 to 7.57]
Statistical Analysis 11: Comparison: 400 mg Moxifloxacin vs Placebo; Comparison at 3.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 6.28, 90% CI 2-sided [3.71 to 8.86]
Statistical Analysis 12: Comparison: 400 mg Moxifloxacin vs Placebo; Comparison at 4.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 6.35, 90% CI 2-sided [3.78 to 8.93]
Statistical Analysis 13: Comparison: 400 mg Moxifloxacin vs Placebo; Comparison at 12.0 hours postdose; Test type: Superiority or Other; LS Mean Difference = 4.71, 90% CI 2-sided [2.11 to 7.31]

ADVERSE EVENTS:
Groups:
- 400 mg Moxifloxican: moxifloxacin: 400 mg tablet, administered orally as a single dose during 1 of 3 treatment periods separated by 2-day washout periods.
Arm/Group | 400 mg LY2140023 | 400 mg Moxifloxican | Placebo
Serious Adverse Events (participants affected / at risk) | 1/81 | 0/82 | 0/80
Other Adverse Events (participants affected / at risk) | 52/81 | 13/82 | 19/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg LY2140023 (N=81) | 400 mg Moxifloxican (N=82) | Placebo (N=80)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg LY2140023 (N=81) | 400 mg Moxifloxican (N=82) | Placebo (N=80)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (18) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (21) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 15 (17) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 4 (4) | 2 (2)
Nystagmus (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days